CLINICAL TRIAL: NCT05537207
Title: Effect of Laser at Lumbar Sensitized Acupoint on Pain Perception and Quality of Life in Female Chronic Pelvic Pain
Brief Title: Laser at Lumbar Acupoint on Pain and Quality of Life in Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/003799
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): low level laser therapy (LLLT) on the acupuncture points.in addition to non-steroidal anti-inflammatory drugs
  Interventions: Device: low level laser therapy; Other: non-steroidal drugs
- control group (Experimental): All women will receive non-steroidal anti-inflammatory drugs in the form of Brufen (Ibuprofen), 400 mg, 3 times per day after meals, for 6 weeks, as will be described by their gynecologist.
  Interventions: Other: non-steroidal drugs

INTERVENTIONS:
Device: low level laser therapy — low level laser therapy (LLLT) on the acupuncture points. inadition to non-steroidal anti-inflammatory drugs.The parameters of the laser device are wave length of 904 nm, maximum average power of 5 milli Watts, a maximum repetition rate of 5 kHz, energy of up to 30 J/cm², and energy density of 2 J/cm2
  Other Names: LLLT
  Arms: study group
Other: non-steroidal drugs — All women will receive non-steroidal anti-inflammatory drugs in the form of Brufen (Ibuprofen), 400 mg, 3 times per day after meals, for 6 weeks, as described by their gynecologist.

SUMMARY:
To investigate the effect of low-level laser at lumbar sensitized acupoint on pain perception in chronic pelvic pain. BACKGROUND: chronic pelvic pain is one of the serious problems in the female, resulting in pain and less physical activity.

DETAILED DESCRIPTION:
Thirty six females with chronic pelvic pain will participate in this study. The patients will randomly be divided into two equal groups; the control group will receive non-steroidal anti-inflammatory drugs in the form of Brufen (Ibuprofen), 400 mg, 3 times per day after meals, for 6 weeks, as will described by their gynecologist. and the study group received the same treatment and low-level laser at lumbar sensitized Acupoint, three times per week for four weeks. The evaluation methods by visual analogue scale (VAS), pain sensitivity was evaluated by measuring mean values of pressure pain thresholds (PPT) using a Pressure Algometer, while the quality of life was evaluated by the 12-Item Short-Form Health Survey (SF-12) before and after the treatment

ELIGIBILITY:
Inclusion Criteria:

* Thirty six female with chronic pelvic pain

  * Their age ranged from 25 to 40 years old.
  * With the maximum parity number three.
  * Their body mass index (BMI) (20:29.9) kg/m2.
  * their pain score on the Visual Analog Scale (VAS) above 4 cm
  * Thirty-six married women diagnosed with chronic pelvic pain (CPP)
  * with a prior history of treatment for pelvic inflammatory disease (PID)
  * women with periodic lower abdominal or pelvic pain for at least six months and met -- the clinical diagnostic criteria for PID based on the presence of all three major criteria: lower abdominal tenderness, cervical motion tenderness, and bilateral adnexal tenderness
  * at least one minor supporting criterion: oral temperature >38.3°C (101 °F), mucopurulent cervical discharge or cervical friability, abundant WBCs on saline microscopy of vaginal fluid, elevated ESR and/or CRP, or laboratory-confirmed cervical infection with N.

gonorrhoeae or C. trachomatis

Exclusion Criteria:

* Any difficulty to communicate or understanding program instructions
* any other conditions that caused pain (for example fibromyalgia and arthritis)
* any psychiatric or cognitive symptoms
* any other musculoskeletal disorders or neurologic diseases
* any other conditions causing pelvic pain (e.g., fibromyalgia, arthritis), history of musculoskeletal or neurological diseases affecting the lower extremities and spine (such as lumbar disc herniation), acute pelvic inflammatory disease (PID), pregnancy or lactation, tumors, pelvic congestion, tuberculous PID, endometriosis, adenomyosis, gynecological tumors, or other gyneco-logical conditions that could contribute to chronic pelvic pain (CPP).
* any issues at acupoint sites (such as ulcers or skin conditions); impairments in other systems that could lead to pelvic and lumbosacral pain (e.g., digestive, motor, or urinary issues)
* severe systemic illnesses affecting the hematologic, digestive, urinary, or cardiovascular systems
* mental illness; cognitive deterioration
* immune-compromising diseases (such as diabetes or HIV/AIDS); and contraindications to NSAIDs

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 4 weeks
  which assesses pain on a paper sheet scale with an increasing number from 0 (no pain) to 10 (the worst pain imaginable).
Pressure Algometer | 4 weeks
  pain sensitivity was evaluated by measuring mean values of pressure pain thresholds (PPT) using a Pressure Algometer. it will be used to assess pain sensitivity through identifying the pressure pain threshold (PPT) for all women before and after treatment. It has a standardized 1.52 cm2 flat circular probe that is pushed against the subject until the pain threshold is reached
Short-Form Health Survey | 4 weeks
  quality of life was evaluated by the 12-Item Short-Form Health Survey (SF-12) before and after the treatment. it is a 12-item questionnaire that was used to assess the quality of life of women in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Lama S Mahmoud, Al Jīzah, Select State, Egypt

REFERENCES:
- [Derived] Hasanin ME, Aly SM, Taha MM, Mahmoud LSE, Aldhahi MI. The Effect of Laser Biostimulation at Sensitized Acupoints on Chronic Pelvic Pain and Quality of Life in Women with Pelvic Inflammatory Disease: A Randomized Controlled Trial. Medicina (Kaunas). 2025 Feb 18;61(2):354. doi: 10.3390/medicina61020354. PMID 40005470